CLINICAL TRIAL: NCT02091401
Title: A Randomized Open-label Study to Compare the Clinical Outcomes and Magnesium Serum Concentrations Obtained in the Treatment of Severe Preeclampsia With a Repeat Bolus Intravenous Magnesium Sulfate Regimen Administered With the Springfusor Infusion Pump to a Continuous Intravenous Magnesium Sulfate Regimen
Brief Title: A Trial Comparing Treatment With the Springfusor Infusion Pump to the IV Magnesium Sulfate Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4002
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Preeclampsia
Keywords: magnesium sulfate
MeSH Terms: conditions — Pre-Eclampsia | interventions — Organization and Administration; Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV (Active Comparator): Women randomized into this treatment group will receive magnesium sulfate via an IV loading dose administered manually by study staff and an IV maintenance regimen.
  Interventions: Other: IV administration; Drug: Magnesium Sulfate
- Springfusor (Experimental): Women randomized into this treatment group will receive magnesium sulfate via IV infusion (with the Springfusor® pump).
  Interventions: Device: Springfusor infusion pump; Drug: Magnesium Sulfate

INTERVENTIONS:
Device: Springfusor infusion pump
  Arms: Springfusor
Other: IV administration
  Arms: IV
Drug: Magnesium Sulfate

SUMMARY:
The trial will test the equivalence of a repeat bolus protocol of magnesium sulfate administered by the Springfusor® controlled pump to a continuous intravenous regimen. The goal of this pharmacokinetic study is to assess the pharmacological equivalence of the serum magnesium sulfate concentrations obtained in the treatment of severe preeclampsia with the continuous intravenous and Springfusor repeat bolus regimens. The study will also document the clinical outcomes, efficacy and acceptability of each treatment for patients and staff.

ELIGIBILITY:
Inclusion Criteria:

Exhibit systolic blood pressure > 160mm Hg OR a diastolic pressure > 110 mm Hg (at two times over 30 minutes) (A single higher pressure could be accepted if the clinical team felt that magnesium sulfate therapy should be initiated without waiting 30 minutes).

Exhibit proteinuria > 1+; Have not given birth, or be <24h postpartum Be assessed by enrolling physician to benefit from magnesium sulfate therapy Agree to comply with study procedures Be > 18 years of age Give informed consent for study participation

Exclusion Criteria:

Eclamptic or seizing at the time of enrollment Received magnesium sulfate therapy 24h prior to study enrollment Known serum creatinine >1.2 mg/dL. (Subject may be enrolled prior to knowledge of serum creatinine but would be withdrawn if >1.2 mg/dL in order to have a proper dose adjustment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Magnesium concentration | 00:00, 00:20; 00:40; 1:20; 2:20; 3:00; 4:40; 5:20; 6:00; 6:20; 7:00; 8:00; 9:40; 10:00; 10:40; 12:00
  Blood draw times will be structured so as to perform a robust population PK analysis. Time zero is the end of the bolus administration. In the Springfusor arm, samples will be collected at the following times: 00:00, 00:20; 00:40; 1:20; 2:00; 2:20; 3:00; 4:40; 5:20; 6:00; 6:20; 7:00; 8:00; 9:40; 10:00; 10:40; 12:00. In the IV arm, samples will be collected at the following times: 0:00; 00:20; 00:40;1:00; 1:20; 1:40; 2:20; 3:00; 3:40; 4:20; 5:20; 6:40; 8:00; 9:20; 10:40 and 12:00.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Bracken, PhD, Study Director — Gynuity Health Projects
Locations (2):
- Egypt (2):
  - Shatby Maternity Hospital, Alexandria
  - El Galaa Teaching Hospital, Cairo

REFERENCES:
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037
- [Derived] Easterling T, Hebert M, Bracken H, Darwish E, Ramadan MC, Shaarawy S, Charles D, Abdel-Aziz T, Nasr AS, Safwal SM, Winikoff B. A randomized trial comparing the pharmacology of magnesium sulfate when used to treat severe preeclampsia with serial intravenous boluses versus a continuous intravenous infusion. BMC Pregnancy Childbirth. 2018 Jul 6;18(1):290. doi: 10.1186/s12884-018-1919-6. PMID 29976161